CLINICAL TRIAL: NCT07109817
Title: Desloratadine to Prevent Taxane-induced Peripheral Neuropathy in Patients With Breast Cancer (DETOXp)
Brief Title: Desloratadine to Prevent Taxane-induced Peripheral Neuropathy in Patients With Breast Cancer
Acronym: DETOXp
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2025-16651
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Peripheral Neuropathy
Keywords: Patient reported outcomes; Biomarkers; Taxane; Neuroinflammatory; Cytokine
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Permuted block randomization procedure will be used for which patients will be randomized between the two treatment arms and stratified using the following criteria specified:
  * Taxane drug: Paclitaxel vs. docetaxel
  * Platinum use: Yes vs. No
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Paclitaxel or Docetaxel for 12 weeks and Placebo
  Interventions: Drug: Placebo
- Desloratodine (Experimental): Paclitaxel or Docetaxel for 12 weeks and Desloratadine
  Interventions: Drug: Desloratodine

INTERVENTIONS:
Drug: Desloratodine — Desloratadine 5mg PO every other day for 12 weeks. Desloratadine is a long- acting tricyclic histamine antagonist with selective H1-receptor histamine antagonist activity. Desloratadine inhibited histamine release from human mast cells.
  Arms: Desloratodine
Drug: Placebo — Placebo daily PO for 12 weeks. Placebo is a lactose filler covered by a capsule.
  Arms: Placebo

SUMMARY:
This is a double-blinded randomized controlled clinical trial that aims to study if desloratadine can reduce rates of peripheral neuropathy development in patients with breast cancer receiving taxane chemotherapy. Researchers will compare desloratadine to a placebo (look-alike substance with no drug) and use validated neurotoxicity and quality of life questionnaires to determine if desloratadine can be used to prevent or make taxane induced peripheral neuropathy (TPIN) symptoms better.

DETAILED DESCRIPTION:
Taxanes are frequently incorporated in first line chemotherapy regimens for breast cancer. Although taxane induces peripheral neuropathy (TIPN) is among the most common side effects of taxane treatment, currently there are no therapies that have consistently proven to be effective in preventing TIPN. TIPN involves a complex interplay of mechanisms which are not yet fully understood. However, neuroinflammation has been shown to be a critical component of the pathophysiology of TIPN. As a result, the discovery of novel therapies that can safely and efficiently attenuate the inflammatory drivers of TIPN and thus prevent the onset of bothersome and potentially disabling neuropathy, represents a unique opportunity to make a meaningful impact on the lives of breast cancer patients.

Desloratadine has shown promise for preventing TIPN in animal models, but based on available information has not yet been tested in humans. This study aims to build on this research by investigating the efficacy of desloratadine in preventing and ameliorating TIPN symptoms as assessed by validated neurotoxicity and quality of life questionnaires. Additionally, this study seeks to expand current knowledge about the role of inflammatory biomarkers as predictive markers of TIPN development. This study will investigate a broad subset of pro and anti-inflammatory cytokines, many of which have been previously shown to be mediated by the Histamine H1 Receptor (HRH1) and 5-HT 2A /c-Fos/NLRP3/IL-1β pathways. This study will measure histamine and nitric oxide levels, which have been show in-vivo to induce neuroinflammation and be upregulated in TIPN. This study will also assess nerve growth factor (NGF) and neurofilament light polypeptide (NF-L), which have protective, regenerative, nociceptive, and structural function in neurons. These biomarkers have shown to correlate with severity of TIPN, but thus far predictive utility is lacking and merits more research. Finally, this study aims to build upon current research regarding the human microbiome and its role in mediating inflammation and the onset of TIPN. Based on current knowledge, no prior study has investigated whether attenuation of chemotherapy induced inflammation via an antihistamine can prevent dysbiosis and help minimize the effect altered gut flora has on promoting further inflammation.

Desloratadine is a safe and inexpensive drug. This study is using 5mg PO dosing, every other day, because this is the standard dose used clinically for allergic rhinitis and chronic urticaria. Based on the effectiveness of loratadine in improving patient reported outcomes from vinca alkaloid induced neuropathy, and because of promising results of desloratadine in preventing and alleviating TIPN in mouse models, it is hypothesized that desloratadine will be an effective therapy to prevent TIPN in patients with breast cancer who receive adjuvant taxane-based chemotherapy regimens. Furthermore, it is also hypothesized that inflammatory biomarkers and gut microbiome signatures are associated with the development of TIPN. The effect of desloratadine in modulating such biomarkers will be monitored.

This double-blinded randomized controlled trial design will help mitigate bias in patient reported outcomes and clinician assessments. If the primary objective is met, desloratadine could potentially represent a safe, cost effective, and accessible strategy to prevent TIPN.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed breast cancer, stage I-III as per the American Joint Committee on Cancer (AJCC) 8th edition (Anatomic Staging)
* Patients must be planned to receive taxane-based regimen for breast cancer (Adjuvant or neoadjuvant) of at least 12 weeks duration. Patients planned to receive taxanes in combination with other chemotherapy drugs (including platinums) are eligible. Patients planned to receive taxanes plus single or dual antiher2 therapy are also eligible. Patients planned to receive taxane-based regimen with immune checkpoint inhibitors are also allowed
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%)
* Patients must have an adequate organ and marrow function as defined below:
* absolute neutrophil count ≥1,000/microliter (mcL)
* platelets ≥100,000/mcL
* total bilirubin ≤ institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
* Creatinine ≤ institutional ULN
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with prior diagnosis of diabetes mellitus are allowed if the patient has no peripheral neuropathy
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants
* Patients must not have received prior taxane or platinum therapy
* Women of childbearing potential must have a negative pregnancy test: serum or urine beta human chorionic gonadotropin (hCG) within 14 days prior to first dose of study treatment
* Potential fertile subjects must agree to use adequate contraception (double barrier methods of birth control or abstinence) prior to start of treatment, for the duration of treatment, and 28 days after last study medication dose. If male, must also agree to refrain from donating sperm during this period

Exclusion Criteria:

* Patients with prior diagnosis of peripheral neuropathy
* Patients who received chemotherapy for the current breast cancer diagnosis before the planned taxane-based regimen
* Patients who are receiving any other investigation agents
* Patients with concurrent use of antihistamines during or for 2 days prior to the study period
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to desloratadine
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant or breastfeeding women are not allowed in the study
* Patients who are taking probiotics
* Patients who are using chronic laxatives or enema
* Patients who used antibiotics within 4 weeks of registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy (FACT)/Gynecologic Oncology Group (GOG)-Neurotoxicity (NTX) Subscale Version 4 (FACT-GOG-NTX) neuropathy score | From baseline to after completion of 12 weeks of taxane chemotherapy
  The patient-related-outcome based neurotoxicity will be assessed using the 11 items about neurotoxicity in the FACT/GOG-NTX questionnaire. For the FACT/GOG-NTX neuropathy, each item is scored from 0-4, and the neurotoxicity total score is the sum of the scores for the 11 items, and ranges from 0 to 44. Lower values of the FACT/GOG-NTX neurotoxicity total score indicate higher neurotoxicity.
  The FACT/GOG-NTX neurotoxicity total score will be analyzed as a continuous variable. Proper transformation to improve normality will be used if needed. Change in FACT/GOG-NTX neuropathy score will be defined as the difference in score values between baseline versus after 12 weeks of taxane chemotherapy.

SECONDARY OUTCOMES:
Rate of grade 2-4 TIPN assessed by treating physician | After completion of 12 weeks of taxane chemotherapy and at 24 weeks and 12 months after completing taxane chemotherapy
  The rate of grade 2-4 TIPN will be assessed by treating physician using CTCAE V5.0 while on taxane treatment. Patients will be coded as having the event if grade 2-4 neuropathy occurred at any time during the observation period. Patients without neuropathy or with maximum of grade 1 neuropathy will be coded as having no event. Of note, only neuropathy with a treatment relationship classified as possibly, probably, or definitely will be considered as taxane-induced neuropathy, whereas neuropathy with a treatment relationship classified as unrelated or unlikely will not be considered an event in the study design.
Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) survey score | After completion of 12 weeks of taxane chemotherapy
  The PRO-CTCAE includes a two-item questionnaire that focuses on taxane-induced peripheral neuropathy (TIPN) in which each item is scored 0 to 4 and a three-item questionnaire that focuses on general pain in which each item is scored 0 to 4. Scores from the two questionnaires are composited yielding an overall possible scoring range of 0-20, such that higher scores represent a patient's self-reported experience of the frequency, severity, and impact of neuropathy and pain on daily activities.
Change in Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT-GOG-NTX) quality of life survey score | From baseline to the completion of 12 weeks of taxane chemotherapy
  The FACT/GOG-NTX quality of life survey score contains 27 questions evaluating 4 domains of quality of life. Each question is scored 0 to 4. The physical wellbeing domain has 7 questions, and the total score ranges from 0-28. The social family well-being domain has 7 questions, and the total score ranges from 0-28. The emotional well-being domain has 6 questions, and the total score ranges from 0-24. The functional well-being score has 7 questions, and the total score ranges from 0-28. The total score for each domain will be summarized and reported as a continuous variable. Researchers will define change in each domain score as the difference in score values between baseline vs. after 12 weeks of taxane chemotherapy.
Change in Patient-Reported Outcomes Measurement Information Systems (PROMIS) 29 v2.1 survey score | From baseline to the completion of 12 weeks of taxane chemotherapy
  The PROMIS 29 survey contains items from seven PROMIS domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities). The PROMIS-29 assesses 7 domains with 4 questions each. There is an additional question that assesses pain intensity 0-10 on numeric rating scale.
  Tables in the protocol will be used to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.
European Organisation of Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) - Chemotherapy-induced Peripheral Neuropathy twenty-item scale (CIPN20) (EORTC QLQ CIPN20) survey score | 12 weeks after the completion of taxane chemotherapy
  The EORTC CIPN20 survey contains 20 items that address neuropathy symptoms using a 4-point Likert type scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"). based on 7-day recall. Given that the patient population in the study is expected to be predominately female and have significant heterogeneity in motor vehicle use, items 19 ("Did you have difficulty using the pedals?") and 20 ("Did you have difficulty getting or maintaining an erection?") will be omitted. The assessment thus can be divided into three subscales: sensory (9 items), motor (7 items), and autonomic symptoms (2 items). Each subscale is converted into a score ranging from 1-36, 1-28, and 1-8, respectively. All scales are linearly converted to a 0-100 total score where a higher score indicates worse symptoms.
Rate of permanent discontinuation of taxane due to TIPN | From baseline up to week 12 of taxane chemotherapy
  The rate of permanent discontinuation of taxane will be calculated as the percentage of patients who discontinue taxane chemotherapy before 12 weeks due to TIPN. Results will be summarized by study arm.
Rate of taxane dose interruption or dose reduction due to TIPN | From baseline up to week 12 of taxane chemotherapy
  The rate of taxane dose interruption or dose reduction will be calculated by the percentage of patients who experience taxane dose interruption or reduction due to TIPN before 12 weeks of taxane treatment. Results will be summarized by study arm.
Rate of pathological complete response (pCR) | After completion of 12 weeks of taxane chemotherapy
  The rate of pathological complete response will be evaluated using the safety of adding desloratadine to taxane-based regimens on breast cancer outcomes. Pathological complete response(pCR), defined as no evidence of invasive carcinoma on breast or axilla after neoadjuvant chemotherapy (ypT0/Tis,ypN0), proposed as a surrogate of overall survival, will be summarized by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus R Anampa, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Giaquinto AN, Jemal A. Cancer statistics, 2024. CA Cancer J Clin. 2024 Jan-Feb;74(1):12-49. doi: 10.3322/caac.21820. Epub 2024 Jan 17. PMID 38230766
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Electronic address: bc.overview@ctsu.ox.ac.uk; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Anthracycline-containing and taxane-containing chemotherapy for early-stage operable breast cancer: a patient-level meta-analysis of 100 000 women from 86 randomised trials. Lancet. 2023 Apr 15;401(10384):1277-1292. doi: 10.1016/S0140-6736(23)00285-4. PMID 37061269
- [Background] Wani MC, Taylor HL, Wall ME, Coggon P, McPhail AT. Plant antitumor agents. VI. The isolation and structure of taxol, a novel antileukemic and antitumor agent from Taxus brevifolia. J Am Chem Soc. 1971 May 5;93(9):2325-7. doi: 10.1021/ja00738a045. No abstract available. PMID 5553076
- [Background] Schiff PB, Fant J, Horwitz SB. Promotion of microtubule assembly in vitro by taxol. Nature. 1979 Feb 22;277(5698):665-7. doi: 10.1038/277665a0. No abstract available. PMID 423966
- [Background] Horwitz SB. Personal recollections on the early development of taxol. J Nat Prod. 2004 Feb;67(2):136-8. doi: 10.1021/np0304464. PMID 14987047
- [Background] Zasadil LM, Andersen KA, Yeum D, Rocque GB, Wilke LG, Tevaarwerk AJ, Raines RT, Burkard ME, Weaver BA. Cytotoxicity of paclitaxel in breast cancer is due to chromosome missegregation on multipolar spindles. Sci Transl Med. 2014 Mar 26;6(229):229ra43. doi: 10.1126/scitranslmed.3007965. PMID 24670687
- [Background] Weaver BA. How Taxol/paclitaxel kills cancer cells. Mol Biol Cell. 2014 Sep 15;25(18):2677-81. doi: 10.1091/mbc.E14-04-0916. PMID 25213191
- [Background] Cortes JE, Pazdur R. Docetaxel. J Clin Oncol. 1995 Oct;13(10):2643-55. doi: 10.1200/JCO.1995.13.10.2643. PMID 7595719
- [Background] Gradishar WJ. Albumin-bound paclitaxel: a next-generation taxane. Expert Opin Pharmacother. 2006 Jun;7(8):1041-53. doi: 10.1517/14656566.7.8.1041. PMID 16722814
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Peto R, Davies C, Godwin J, Gray R, Pan HC, Clarke M, Cutter D, Darby S, McGale P, Taylor C, Wang YC, Bergh J, Di Leo A, Albain K, Swain S, Piccart M, Pritchard K. Comparisons between different polychemotherapy regimens for early breast cancer: meta-analyses of long-term outcome among 100,000 women in 123 randomised trials. Lancet. 2012 Feb 4;379(9814):432-44. doi: 10.1016/S0140-6736(11)61625-5. Epub 2011 Dec 5. PMID 22152853
- [Background] Rowinsky EK, Donehower RC. Paclitaxel (taxol). N Engl J Med. 1995 Apr 13;332(15):1004-14. doi: 10.1056/NEJM199504133321507. No abstract available. PMID 7885406
- [Background] Ringel I, Horwitz SB. Studies with RP 56976 (taxotere): a semisynthetic analogue of taxol. J Natl Cancer Inst. 1991 Feb 20;83(4):288-91. doi: 10.1093/jnci/83.4.288. PMID 1671606
- [Background] Schneider BP, Shen F, Jiang G, O'Neill A, Radovich M, Li L, Gardner L, Lai D, Foroud T, Sparano JA, Sledge GW Jr, Miller KD. Impact of Genetic Ancestry on Outcomes in ECOG-ACRIN-E5103. JCO Precis Oncol. 2017;2017:PO.17.00059. doi: 10.1200/PO.17.00059. Epub 2017 Aug 21. PMID 29333527
- [Background] Michalova Z, Szekiova E, Blasko J, Vanicky I. Prevention and therapy of chemotherapy-induced peripheral neuropathy: a review of recent findings. Neoplasma. 2023 Feb;70(1):15-35. doi: 10.4149/neo_2022_221007N992. Epub 2022 Dec 28. PMID 36573482
- [Background] Sahenk Z, Barohn R, New P, Mendell JR. Taxol neuropathy. Electrodiagnostic and sural nerve biopsy findings. Arch Neurol. 1994 Jul;51(7):726-9. doi: 10.1001/archneur.1994.00540190110024. PMID 7912506
- [Background] Komiya Y, Tashiro T. Effects of taxol on slow and fast axonal transport. Cell Motil Cytoskeleton. 1988;11(3):151-6. doi: 10.1002/cm.970110302. PMID 2463106
- [Background] Han Y, Smith MT. Pathobiology of cancer chemotherapy-induced peripheral neuropathy (CIPN). Front Pharmacol. 2013 Dec 18;4:156. doi: 10.3389/fphar.2013.00156. PMID 24385965
- [Background] Guo C, Sun L, Chen X, Zhang D. Oxidative stress, mitochondrial damage and neurodegenerative diseases. Neural Regen Res. 2013 Jul 25;8(21):2003-14. doi: 10.3969/j.issn.1673-5374.2013.21.009. PMID 25206509
- [Background] Zhang H, Boyette-Davis JA, Kosturakis AK, Li Y, Yoon SY, Walters ET, Dougherty PM. Induction of monocyte chemoattractant protein-1 (MCP-1) and its receptor CCR2 in primary sensory neurons contributes to paclitaxel-induced peripheral neuropathy. J Pain. 2013 Oct;14(10):1031-44. doi: 10.1016/j.jpain.2013.03.012. Epub 2013 May 31. PMID 23726937
- [Background] Binshtok AM, Wang H, Zimmermann K, Amaya F, Vardeh D, Shi L, Brenner GJ, Ji RR, Bean BP, Woolf CJ, Samad TA. Nociceptors are interleukin-1beta sensors. J Neurosci. 2008 Dec 24;28(52):14062-73. doi: 10.1523/JNEUROSCI.3795-08.2008. PMID 19109489
- [Background] Sorkin LS, Xiao WH, Wagner R, Myers RR. Tumour necrosis factor-alpha induces ectopic activity in nociceptive primary afferent fibres. Neuroscience. 1997 Nov;81(1):255-62. doi: 10.1016/s0306-4522(97)00147-4. PMID 9300418
- [Background] Ozaktay AC, Cavanaugh JM, Asik I, DeLeo JA, Weinstein JN. Dorsal root sensitivity to interleukin-1 beta, interleukin-6 and tumor necrosis factor in rats. Eur Spine J. 2002 Oct;11(5):467-75. doi: 10.1007/s00586-002-0430-x. Epub 2002 Jun 4. PMID 12384756
- [Background] McMahon SB, Cafferty WB, Marchand F. Immune and glial cell factors as pain mediators and modulators. Exp Neurol. 2005 Apr;192(2):444-62. doi: 10.1016/j.expneurol.2004.11.001. PMID 15755561
- [Background] Loprinzi CL, Lacchetti C, Bleeker J, Cavaletti G, Chauhan C, Hertz DL, Kelley MR, Lavino A, Lustberg MB, Paice JA, Schneider BP, Lavoie Smith EM, Smith ML, Smith TJ, Wagner-Johnston N, Hershman DL. Prevention and Management of Chemotherapy-Induced Peripheral Neuropathy in Survivors of Adult Cancers: ASCO Guideline Update. J Clin Oncol. 2020 Oct 1;38(28):3325-3348. doi: 10.1200/JCO.20.01399. Epub 2020 Jul 14. PMID 32663120
- [Background] Huang HQ, Brady MF, Cella D, Fleming G. Validation and reduction of FACT/GOG-Ntx subscale for platinum/paclitaxel-induced neurologic symptoms: a gynecologic oncology group study. Int J Gynecol Cancer. 2007 Mar-Apr;17(2):387-93. doi: 10.1111/j.1525-1438.2007.00794.x. PMID 17362317
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Cheng HL, Lopez V, Lam SC, Leung AKT, Li YC, Wong KH, Au JSK, Sundar R, Chan A, De Ng TR, Suen LKP, Chan CW, Yorke J, Molassiotis A. Psychometric testing of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) subscale in a longitudinal study of cancer patients treated with chemotherapy. Health Qual Life Outcomes. 2020 Jul 23;18(1):246. doi: 10.1186/s12955-020-01493-y. PMID 32703223
- [Background] Beijers AJM, Bonhof CS, Mols F, Ophorst J, de Vos-Geelen J, Jacobs EMG, van de Poll-Franse LV, Vreugdenhil G. Multicenter randomized controlled trial to evaluate the efficacy and tolerability of frozen gloves for the prevention of chemotherapy-induced peripheral neuropathy. Ann Oncol. 2020 Jan;31(1):131-136. doi: 10.1016/j.annonc.2019.09.006. PMID 31912787
- [Background] Norman GR, Sloan JA, Wyrwich KW. Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. Med Care. 2003 May;41(5):582-92. doi: 10.1097/01.MLR.0000062554.74615.4C. PMID 12719681
- [Background] Tsuyuki S, Yamagami K, Yoshibayashi H, Sugie T, Mizuno Y, Tanaka S, Kato H, Okuno T, Ogura N, Yamashiro H, Takuwa H, Kikawa Y, Hashimoto T, Kato T, Takahara S, Katayama T, Yamauchi A, Inamoto T. Effectiveness and safety of surgical glove compression therapy as a prophylactic method against nanoparticle albumin-bound-paclitaxel-induced peripheral neuropathy. Breast. 2019 Oct;47:22-27. doi: 10.1016/j.breast.2019.06.008. Epub 2019 Jul 3. PMID 31302389
- [Background] Su Y, Huang J, Wang S, Unger JM, Arias-Fuenzalida J, Shi Y, Li J, Gao Y, Shi W, Wang X, Peng R, Xu F, An X, Xue C, Xia W, Hong R, Zhong Y, Lin Y, Huang H, Zhang A, Zhang L, Cai L, Zhang J, Yuan Z. The Effects of Ganglioside-Monosialic Acid in Taxane-Induced Peripheral Neurotoxicity in Patients with Breast Cancer: A Randomized Trial. J Natl Cancer Inst. 2020 Jan 1;112(1):55-62. doi: 10.1093/jnci/djz086. PMID 31093677
- [Background] Murdoch D, Goa KL, Keam SJ. Desloratadine: an update of its efficacy in the management of allergic disorders. Drugs. 2003;63(19):2051-77. doi: 10.2165/00003495-200363190-00010. PMID 12962522
- [Background] Anampa J, Makower D, Sparano JA. Progress in adjuvant chemotherapy for breast cancer: an overview. BMC Med. 2015 Aug 17;13:195. doi: 10.1186/s12916-015-0439-8. PMID 26278220
- [Background] Liu X, Tonello R, Ling Y, Gao YJ, Berta T. Paclitaxel-activated astrocytes produce mechanical allodynia in mice by releasing tumor necrosis factor-alpha and stromal-derived cell factor 1. J Neuroinflammation. 2019 Nov 10;16(1):209. doi: 10.1186/s12974-019-1619-9. PMID 31707979
- [Background] Brandolini L, d'Angelo M, Novelli R, Castelli V, Giorgio C, Sirico A, Cocchiaro P, D'Egidio F, Benedetti E, Cristiano C, Bugatti A, Ruocco A, Amendola PG, Talarico C, Manelfi C, Iaconis D, Beccari A, Quadros AU, Cunha TM, Caruso A, Russo R, Cimini A, Aramini A, Allegretti M. Paclitaxel binds and activates C5aR1: A new potential therapeutic target for the prevention of chemotherapy-induced peripheral neuropathy and hypersensitivity reactions. Cell Death Dis. 2022 May 25;13(5):500. doi: 10.1038/s41419-022-04964-w. PMID 35614037
- [Background] Escribese MM, Rosace D, Chivato T, Fernandez TD, Corbi AL, Barber D. Alternative Anaphylactic Routes: The Potential Role of Macrophages. Front Immunol. 2017 May 8;8:515. doi: 10.3389/fimmu.2017.00515. eCollection 2017. PMID 28533777
- [Background] Wang J, Zhou Y, Zhang H, Hu L, Liu J, Wang L, Wang T, Zhang H, Cong L, Wang Q. Pathogenesis of allergic diseases and implications for therapeutic interventions. Signal Transduct Target Ther. 2023 Mar 24;8(1):138. doi: 10.1038/s41392-023-01344-4. PMID 36964157
- [Background] Yu J, Lou GD, Yue JX, Tang YY, Hou WW, Shou WT, Ohtsu H, Zhang SH, Chen Z. Effects of histamine on spontaneous neuropathic pain induced by peripheral axotomy. Neurosci Bull. 2013 Jun;29(3):261-9. doi: 10.1007/s12264-013-1316-0. Epub 2013 Mar 13. PMID 23494529
- [Background] Hunto ST, Kim HG, Baek KS, Jeong D, Kim E, Kim JH, Cho JY. Loratadine, an antihistamine drug, exhibits anti-inflammatory activity through suppression of the NF-kB pathway. Biochem Pharmacol. 2020 Jul;177:113949. doi: 10.1016/j.bcp.2020.113949. Epub 2020 Apr 3. PMID 32251678
- [Background] Jang J, Hunto ST, Kim JW, Lee HP, Kim HG, Cho JY. Anti-Inflammatory Activities of an Anti-Histamine Drug, Loratadine, by Suppressing TAK1 in AP-1 Pathway. Int J Mol Sci. 2022 Apr 3;23(7):3986. doi: 10.3390/ijms23073986. PMID 35409346
- [Background] Kamal N, Abdallah MS, Abdel Wahed E, Sabri NA, Fahmy SF. Evaluation of the Effect of Loratadine versus Diosmin/Hesperidin Combination on Vinca Alkaloids-Induced Neuropathy: A Randomized Controlled Clinical Trial. Pharmaceuticals (Basel). 2024 May 9;17(5):609. doi: 10.3390/ph17050609. PMID 38794179
- [Background] Canonica GW, Blaiss M. Antihistaminic, anti-inflammatory, and antiallergic properties of the nonsedating second-generation antihistamine desloratadine: a review of the evidence. World Allergy Organ J. 2011 Feb;4(2):47-53. doi: 10.1097/WOX.0b013e3182093e19. Epub 2011 Feb 23. PMID 23268457
- [Background] Wu RL, Anthes JC, Kreutner W, Harris AG, West RE Jr. Desloratadine inhibits constitutive and histamine-stimulated nuclear factor-kappaB activity consistent with inverse agonism at the histamine H1 Receptor. Int Arch Allergy Immunol. 2004 Dec;135(4):313-8. doi: 10.1159/000082325. Epub 2004 Nov 24. PMID 15564772
- [Background] Lu J, Zhao XJ, Ruan Y, Liu XJ, Di X, Xu R, Wang JY, Qian MY, Jin HM, Li WJ, Shen X. Desloratadine ameliorates paclitaxel-induced peripheral neuropathy and hypersensitivity reactions in mice. Acta Pharmacol Sin. 2024 Oct;45(10):2061-2076. doi: 10.1038/s41401-024-01301-z. Epub 2024 May 24. PMID 38789495
- [Background] Ma J, Kavelaars A, Dougherty PM, Heijnen CJ. Beyond symptomatic relief for chemotherapy-induced peripheral neuropathy: Targeting the source. Cancer. 2018 Jun 1;124(11):2289-2298. doi: 10.1002/cncr.31248. Epub 2018 Feb 20. PMID 29461625
- [Background] Boyette-Davis JA, Cata JP, Driver LC, Novy DM, Bruel BM, Mooring DL, Wendelschafer-Crabb G, Kennedy WR, Dougherty PM. Persistent chemoneuropathy in patients receiving the plant alkaloids paclitaxel and vincristine. Cancer Chemother Pharmacol. 2013 Mar;71(3):619-26. doi: 10.1007/s00280-012-2047-z. Epub 2012 Dec 11. PMID 23228992
- [Background] Aloe L, Rocco ML, Bianchi P, Manni L. Nerve growth factor: from the early discoveries to the potential clinical use. J Transl Med. 2012 Nov 29;10:239. doi: 10.1186/1479-5876-10-239. PMID 23190582
- [Background] Cavaletti G, Bogliun G, Marzorati L, Zincone A, Piatti M, Colombo N, Franchi D, La Presa MT, Lissoni A, Buda A, Fei F, Cundari S, Zanna C. Early predictors of peripheral neurotoxicity in cisplatin and paclitaxel combination chemotherapy. Ann Oncol. 2004 Sep;15(9):1439-42. doi: 10.1093/annonc/mdh348. PMID 15319252
- [Background] Rodwin RL, Siddiq NZ, Ehrlich BE, Lustberg MB. Biomarkers of Chemotherapy-Induced Peripheral Neuropathy: Current Status and Future Directions. Front Pain Res (Lausanne). 2022 Mar 14;3:864910. doi: 10.3389/fpain.2022.864910. eCollection 2022. PMID 35360655
- [Background] Karteri S, Bruna J, Argyriou AA, Mariotto S, Velasco R, Alemany M, Kalofonou F, Alberti P, Dinoto A, Velissaris D, Stradella A, Cavaletti G, Ferrari S, Kalofonos HP. Prospectively assessing serum neurofilament light chain levels as a biomarker of paclitaxel-induced peripheral neurotoxicity in breast cancer patients. J Peripher Nerv Syst. 2022 Jun;27(2):166-174. doi: 10.1111/jns.12493. Epub 2022 Apr 13. PMID 35384143
- [Background] Youk J, Kim YS, Lim JA, Shin DY, Koh Y, Lee ST, Kim I. Depletion of nerve growth factor in chemotherapy-induced peripheral neuropathy associated with hematologic malignancies. PLoS One. 2017 Aug 21;12(8):e0183491. doi: 10.1371/journal.pone.0183491. eCollection 2017. PMID 28827818
- [Background] Shatunova S, Aktar R, Peiris M, Lee JYP, Vetter I, Starobova H. The role of the gut microbiome in neuroinflammation and chemotherapy-induced peripheral neuropathy. Eur J Pharmacol. 2024 Sep 15;979:176818. doi: 10.1016/j.ejphar.2024.176818. Epub 2024 Jul 18. PMID 39029779
- [Background] Singh SK, Krukowski K, Laumet GO, Weis D, Alexander JF, Heijnen CJ, Kavelaars A. CD8+ T cell-derived IL-13 increases macrophage IL-10 to resolve neuropathic pain. JCI Insight. 2022 Mar 8;7(5):e154194. doi: 10.1172/jci.insight.154194. PMID 35260535
- [Background] Uceyler N, Rogausch JP, Toyka KV, Sommer C. Differential expression of cytokines in painful and painless neuropathies. Neurology. 2007 Jul 3;69(1):42-9. doi: 10.1212/01.wnl.0000265062.92340.a5. PMID 17606879
- [Background] Kleckner IR, Jusko TA, Culakova E, Chung K, Kleckner AS, Asare M, Inglis JE, Loh KP, Peppone LJ, Miller J, Melnik M, Kasbari S, Ossip D, Mustian KM. Longitudinal study of inflammatory, behavioral, clinical, and psychosocial risk factors for chemotherapy-induced peripheral neuropathy. Breast Cancer Res Treat. 2021 Sep;189(2):521-532. doi: 10.1007/s10549-021-06304-6. Epub 2021 Jun 30. PMID 34191201
- [Background] Rumore MM, Schlichting DA. Clinical efficacy of antihistaminics as analgesics. Pain. 1986 Apr;25(1):7-22. doi: 10.1016/0304-3959(86)90004-7. PMID 2872645
- [Background] Al-Mazidi S, Alotaibi M, Nedjadi T, Chaudhary A, Alzoghaibi M, Djouhri L. Blocking of cytokines signalling attenuates evoked and spontaneous neuropathic pain behaviours in the paclitaxel rat model of chemotherapy-induced neuropathy. Eur J Pain. 2018 Apr;22(4):810-821. doi: 10.1002/ejp.1169. Epub 2017 Dec 27. PMID 29282807
- [Background] Manjavachi MN, Passos GF, Trevisan G, Araujo SB, Pontes JP, Fernandes ES, Costa R, Calixto JB. Spinal blockage of CXCL1 and its receptor CXCR2 inhibits paclitaxel-induced peripheral neuropathy in mice. Neuropharmacology. 2019 Jun;151:136-143. doi: 10.1016/j.neuropharm.2019.04.014. Epub 2019 Apr 13. PMID 30991054
- [Background] Nakamura T, Kawarabayashi T, Shibata M, Kasahara H, Makioka K, Sugawara T, Oka H, Ishizawa K, Amari M, Ueda T, Kinoshita S, Miyamoto Y, Kaito K, Takatama M, Ikeda Y, Shoji M. High levels of plasma neurofilament light chain correlated with brainstem and peripheral nerve damage. J Neurol Sci. 2024 Aug 15;463:123137. doi: 10.1016/j.jns.2024.123137. Epub 2024 Jul 15. PMID 39032446
- [Background] Velasco R, Marco C, Domingo-Domenech E, Stradella A, Santos C, Laquente B, Ferrer G, Argyriou AA, Bruna J. Plasma neurofilament light chain levels in chemotherapy-induced peripheral neurotoxicity according to type of anticancer drug. Eur J Neurol. 2024 Sep;31(9):e16369. doi: 10.1111/ene.16369. Epub 2024 Jul 1. PMID 38952074
- [Background] Furman D, Campisi J, Verdin E, Carrera-Bastos P, Targ S, Franceschi C, Ferrucci L, Gilroy DW, Fasano A, Miller GW, Miller AH, Mantovani A, Weyand CM, Barzilai N, Goronzy JJ, Rando TA, Effros RB, Lucia A, Kleinstreuer N, Slavich GM. Chronic inflammation in the etiology of disease across the life span. Nat Med. 2019 Dec;25(12):1822-1832. doi: 10.1038/s41591-019-0675-0. Epub 2019 Dec 5. PMID 31806905
- [Background] Muller DN, Wilck N, Haase S, Kleinewietfeld M, Linker RA. Sodium in the microenvironment regulates immune responses and tissue homeostasis. Nat Rev Immunol. 2019 Apr;19(4):243-254. doi: 10.1038/s41577-018-0113-4. PMID 30644452
- [Background] Chassaing B, Van de Wiele T, De Bodt J, Marzorati M, Gewirtz AT. Dietary emulsifiers directly alter human microbiota composition and gene expression ex vivo potentiating intestinal inflammation. Gut. 2017 Aug;66(8):1414-1427. doi: 10.1136/gutjnl-2016-313099. Epub 2017 Mar 21. PMID 28325746
- [Background] Meneses-Echavez JF, Correa-Bautista JE, Gonzalez-Jimenez E, Schmidt Rio-Valle J, Elkins MR, Lobelo F, Ramirez-Velez R. The Effect of Exercise Training on Mediators of Inflammation in Breast Cancer Survivors: A Systematic Review with Meta-analysis. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1009-17. doi: 10.1158/1055-9965.EPI-15-1061. Epub 2016 Apr 12. PMID 27197276
- [Background] Khanna D, Khanna S, Khanna P, Kahar P, Patel BM. Obesity: A Chronic Low-Grade Inflammation and Its Markers. Cureus. 2022 Feb 28;14(2):e22711. doi: 10.7759/cureus.22711. eCollection 2022 Feb. PMID 35386146
- [Background] Reutrakul S, Van Cauter E. Sleep influences on obesity, insulin resistance, and risk of type 2 diabetes. Metabolism. 2018 Jul;84:56-66. doi: 10.1016/j.metabol.2018.02.010. Epub 2018 Mar 3. PMID 29510179
- [Background] Cohen S, Janicki-Deverts D, Doyle WJ, Miller GE, Frank E, Rabin BS, Turner RB. Chronic stress, glucocorticoid receptor resistance, inflammation, and disease risk. Proc Natl Acad Sci U S A. 2012 Apr 17;109(16):5995-9. doi: 10.1073/pnas.1118355109. Epub 2012 Apr 2. PMID 22474371
- [Background] Ghoreishi Z, Keshavarz S, Asghari Jafarabadi M, Fathifar Z, Goodman KA, Esfahani A. Risk factors for paclitaxel-induced peripheral neuropathy in patients with breast cancer. BMC Cancer. 2018 Oct 5;18(1):958. doi: 10.1186/s12885-018-4869-5. PMID 30290775
- [Background] Greenlee H, Hershman DL, Shi Z, Kwan ML, Ergas IJ, Roh JM, Kushi LH. BMI, Lifestyle Factors and Taxane-Induced Neuropathy in Breast Cancer Patients: The Pathways Study. J Natl Cancer Inst. 2016 Oct 28;109(2):djw206. doi: 10.1093/jnci/djw206. Print 2017 Feb. PMID 27794123
- [Background] Zhang F, Aschenbrenner D, Yoo JY, Zuo T. The gut mycobiome in health, disease, and clinical applications in association with the gut bacterial microbiome assembly. Lancet Microbe. 2022 Dec;3(12):e969-e983. doi: 10.1016/S2666-5247(22)00203-8. Epub 2022 Sep 28. PMID 36182668
- [Background] Otto-Dobos LD, Grant CV, Lahoud AA, Wilcox OR, Strehle LD, Loman BR, Adarkwah Yiadom S, Seng MM, Halloy NR, Russart KLG, Carpenter KM, Dawson E, Sardesai SD, Williams NO, Gatti-Mays ME, Stover DG, Sudheendra PK, Wesolowski R, Kiecolt-Glaser JK, Bailey MT, Andridge RR, Pyter LM. Chemotherapy-induced gut microbiome disruption, inflammation, and cognitive decline in female patients with breast cancer. Brain Behav Immun. 2024 Aug;120:208-220. doi: 10.1016/j.bbi.2024.05.039. Epub 2024 May 31. PMID 38823430
- [Background] Ramakrishna C, Corleto J, Ruegger PM, Logan GD, Peacock BB, Mendonca S, Yamaki S, Adamson T, Ermel R, McKemy D, Borneman J, Cantin EM. Dominant Role of the Gut Microbiota in Chemotherapy Induced Neuropathic Pain. Sci Rep. 2019 Dec 30;9(1):20324. doi: 10.1038/s41598-019-56832-x. PMID 31889131
- [Background] Cuozzo M, Castelli V, Avagliano C, Cimini A, d'Angelo M, Cristiano C, Russo R. Effects of Chronic Oral Probiotic Treatment in Paclitaxel-Induced Neuropathic Pain. Biomedicines. 2021 Mar 30;9(4):346. doi: 10.3390/biomedicines9040346. PMID 33808052
- [Background] Shen S, Lim G, You Z, Ding W, Huang P, Ran C, Doheny J, Caravan P, Tate S, Hu K, Kim H, McCabe M, Huang B, Xie Z, Kwon D, Chen L, Mao J. Gut microbiota is critical for the induction of chemotherapy-induced pain. Nat Neurosci. 2017 Sep;20(9):1213-1216. doi: 10.1038/nn.4606. Epub 2017 Jul 17. PMID 28714953
- [Background] Terrisse S, Derosa L, Iebba V, Ghiringhelli F, Vaz-Luis I, Kroemer G, Fidelle M, Christodoulidis S, Segata N, Thomas AM, Martin AL, Sirven A, Everhard S, Aprahamian F, Nirmalathasan N, Aarnoutse R, Smidt M, Ziemons J, Caldas C, Loibl S, Denkert C, Durand S, Iglesias C, Pietrantonio F, Routy B, Andre F, Pasolli E, Delaloge S, Zitvogel L. Intestinal microbiota influences clinical outcome and side effects of early breast cancer treatment. Cell Death Differ. 2021 Sep;28(9):2778-2796. doi: 10.1038/s41418-021-00784-1. Epub 2021 May 7. PMID 33963313
- [Background] Lavoie Smith EM, Barton DL, Qin R, Steen PD, Aaronson NK, Loprinzi CL. Assessing patient-reported peripheral neuropathy: the reliability and validity of the European Organization for Research and Treatment of Cancer QLQ-CIPN20 Questionnaire. Qual Life Res. 2013 Dec;22(10):2787-99. doi: 10.1007/s11136-013-0379-8. Epub 2013 Mar 30. PMID 23543373
- [Background] Le-Rademacher J, Kanwar R, Seisler D, Pachman DR, Qin R, Abyzov A, Ruddy KJ, Banck MS, Lavoie Smith EM, Dorsey SG, Aaronson NK, Sloan J, Loprinzi CL, Beutler AS. Patient-reported (EORTC QLQ-CIPN20) versus physician-reported (CTCAE) quantification of oxaliplatin- and paclitaxel/carboplatin-induced peripheral neuropathy in NCCTG/Alliance clinical trials. Support Care Cancer. 2017 Nov;25(11):3537-3544. doi: 10.1007/s00520-017-3780-y. Epub 2017 Jun 20. PMID 28634656
- [Background] Calhoun EA, Welshman EE, Chang CH, Lurain JR, Fishman DA, Hunt TL, Cella D. Psychometric evaluation of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (Fact/GOG-Ntx) questionnaire for patients receiving systemic chemotherapy. Int J Gynecol Cancer. 2003 Nov-Dec;13(6):741-8. doi: 10.1111/j.1525-1438.2003.13603.x. PMID 14675309
- [Background] Cella D, Peterman A, Hudgens S, Webster K, Socinski MA. Measuring the side effects of taxane therapy in oncology: the functional assesment of cancer therapy-taxane (FACT-taxane). Cancer. 2003 Aug 15;98(4):822-31. doi: 10.1002/cncr.11578. PMID 12910528
- [Background] Hershman DL, Unger JM, Crew KD, Minasian LM, Awad D, Moinpour CM, Hansen L, Lew DL, Greenlee H, Fehrenbacher L, Wade JL 3rd, Wong SF, Hortobagyi GN, Meyskens FL, Albain KS. Randomized double-blind placebo-controlled trial of acetyl-L-carnitine for the prevention of taxane-induced neuropathy in women undergoing adjuvant breast cancer therapy. J Clin Oncol. 2013 Jul 10;31(20):2627-33. doi: 10.1200/JCO.2012.44.8738. Epub 2013 Jun 3. PMID 23733756
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J. The Functional Assessment of Cancer Therapy Scale: Development and Validation of the General Measure. J Clin Oncol. 2023 Dec 10;41(35):5335-5344. doi: 10.1200/JCO.22.02775. PMID 38056080
- [Background] Park SB, Goldstein D, Krishnan AV, Lin CS, Friedlander ML, Cassidy J, Koltzenburg M, Kiernan MC. Chemotherapy-induced peripheral neurotoxicity: a critical analysis. CA Cancer J Clin. 2013 Nov-Dec;63(6):419-37. doi: 10.3322/caac.21204. PMID 24590861